CLINICAL TRIAL: NCT05822193
Title: Incidence, Associated Factors, and Burden of Post COVID-19 Condition in Brazil
Status: Recruiting | Type: Observational
Sponsor: Inova Medical (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023/001
Record Dates: First submitted 2023-04-18; First posted 2023-04-20 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Post-Acute COVID-19 Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Individuals with COVID-19 diagnosis during the SARS-CoV-2 omicron wave in Brazil
  Interventions: Other: Multiple exposures

INTERVENTIONS:
Other: Multiple exposures — Exposures variables (observational study): age, gender, education, comorbidities, vaccination status, severity of the acute episode of COVID-19, treatments used for acute COVID-19.

SUMMARY:
This is a national retrospective cohort study with internet-based recruitment which intends to enroll 1,694 adult patients with COVID-19 diagnosis during the SARS-CoV-2 omicron wave in Brazil. Participants with confirmed symptomatic COVID-19 after january 2022 will be evaluated in order to assess incidence, potential risk factors and impact of post COVID-19 condition according to the WHO definition on health-related quality of life and other relevant patient-centered outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Brazilian resident;
* Symptomatica COVID-19 confirmed by reverse transcriptase polymerase chain reaction (RT-PCR) or antigen test for SARS-COV-2 after January 2022, with diagnosis at least 90 days before recruitment.

Exclusion Criteria:

* No availability to participate in remote research appointments;
* Communication difficulty (aphasia, important hearing loss, non-portuguese speaker, severe dementia)
* Refuse to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study target population is composed by adult participants with confirmed symptomatic COVID-19 during the SARS-CoV-2 omicron wave in Brazil (January 2022 to date, representing the period of time with absolute dominance of omicron as circulating variant). The study will include patients with distinct levels of acute illness severity (i.e., both outpatients and patients who required hospitalization for COVID-19).
Sampling Method: Non-Probability Sample
Enrollment: 1694 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Post COVID-19 condition according to the WHO definition | 3 to 24 months
  Post COVID-19 condition occurs in individuals with a history of probable or confirmed SARS CoV-2 infection, usually 3 months from the onset of COVID-19 with symptoms and that last for at least 2 months and cannot be explained by an alternative diagnosis
EQ5D-3L | 3 to 24 months
  Health-related quality of life assessed using the EuroQol five-dimensional 3-level descriptive system (EQ5D-3L). This outcome will be considered as primary when Post COVID-19 condition be used as exposure.

SECONDARY OUTCOMES:
Instrumental activities of daily living | 3 to 24 months
  Instrumental activities of daily living assessed with the Lawton & Brody Instrumental Activities of Daily Living
Functional status | 3 to 24 months
  Functional status assessed with the Modified Barthel Index
Cognition | 3 to 24 months
  Cognition assessed with the Telephone Interview for Cognitive Status
Anxiety symptoms | 3 to 24 months
  Anxiety symptoms assessed with the Hospital Anxiety and Depression Scale;
Depression symptoms | 3 to 24 months
  Depression symptoms assessed with the Hospital Anxiety and Depression Scale;
Posttraumatic stress symptoms | 3 to 24 months
  Posttraumatic stress symptoms assessed with the Impact Event Scale-Revised
Time to return to work or studies | 3 to 24 months
  Time to return to work or studies after COVID-19
Healthcare utilization | 3 to 24 months
  Medical and rehabilitation appointments, medication use and diagnostic tests
Costs | 3 to 24 months
  Individual health-related and COVID-19-related costs

CONTACTS AND LOCATIONS:
Locations (1):
- Inova Medical, Cachoeirinha, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
To be disclosed